CLINICAL TRIAL: NCT02888288
Title: Integrating Mental Health Into a HIV Clinic to Improve Outcomes Among Tanzanian Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00069892
Record Dates: First submitted 2016-08-09; First posted 2016-09-05 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Health Behavior; HIV; Mental Health
Keywords: adolescent; adolescence; HIV/AIDS; mental health; cognitive behavioral therapy
MeSH Terms: conditions — Health Behavior; Psychological Well-Being; Acquired Immunodeficiency Syndrome | interventions — Play Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mental Health Intervention (Experimental): This arm was designed based on mental health needs of HIV-infected youth in Tanzania. It incorporates principles of cognitive behavioral therapy, interpersonal psychotherapy, and motivational interviewing built into 10 group sessions, approximately 90 minutes each (2 sessions with caregiver participation) and 2 individual sessions. Groups are age and gender matched and facilitated by lay counselors with a mix of lived experience and prior mental health research experience.
  Interventions: Behavioral: Mental Health Intervention
- Standard of Care (Active Comparator): This arm includes standard medical care and adherence counseling with routine education prior to the start of the HIV youth clinic from which participants are recruited.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Mental Health Intervention — Includes a standard format of greetings, review of last session content, homework discussion, new topic, assigning homework and ends with a fun activity, relaxation or game. First session is a joint session with youth and caregivers. Topics include common stresses and worries experienced by HIV+ youth; relaxation and coping techniques; cognitive behavioral triangle; story of finding out HIV status and if willing, to discuss this in an individual session, peer group session, and with caregiver; identify circles of support; discuss stigma and how to disclose HIV status to others; consider values, hopes and dreams for the future, and how to use this information to live positively with HIV. ART adherence is woven into case examples and discussions.
  Arms: Mental Health Intervention
Behavioral: Standard of Care — Standard of Care includes enhanced ART adherence based on clinic protocols and monthly HIV teaching sessions prior to adolescent clinic.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate if a group-based mental health intervention called Sauti ya Vijana (The Voice of Youth) designed to address mental health challenges faced by adolescents in Tanzania is acceptable and feasible and if it improves mental health, antiretroviral therapy (ART) adherence, and virologic outcomes among HIV-positive adolescents as compared to youth receiving treatment as usual. Mental health intervention sessions will take place three times a month for approximately four months in groups of eight to ten youth based on age and sex. Caregivers will attend two sessions to support the youth and provide the guardian perspective on caring for HIV-positive adolescents. The investigator hypothesizes the mental health intervention will be acceptable, feasible, and will improve mental health and ART adherence among participating youth and this improvement will be sustained over time.

DETAILED DESCRIPTION:
The study will enroll up to approximately 130 participants from the established Kilimanjaro Christian Medical Centre and Mawenzi Saturday Teen Clinics. Participants will be assigned to approximately eight to ten persons per group, based on age and sex. Groups will be matched in pairs as closely as possible (ex. two groups of females 12-16 years of age) and assigned to Wave 1, 2, or 3. Randomization will occur on the individual level and will occur just before the start of mental health intervention for each wave. Individuals will be randomized at this time point to reduce potential drop out of those with delayed start (Wave 2/3). Randomization will occur by a coin flip for two individuals based on alphabetical order: heads will be intervention group (I) and tails the standard of care group (SOC).

This feasibility study is longitudinal with up to 24 month follow-up after intervention. Feasibility measures from lay counselors will be monitored weekly. Outcome measures will be obtained by blinded interviewers using a structured survey to inquire about mental health symptoms, self-report adherence, obtain an ART drug concentration level from a hair sample, and HIV-1 viral load from a blood sample and will be collected by the same research assistants at five to six potential time points: 1) baseline, 2) pre-intervention, 3) post-intervention, 4) 6-months post-intervention, 5) 12-months post-intervention and 6) 24-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Youth between the ages of 12 and 24 years of age, attending the Teen Club HIV clinic at Kilimanjaro Christian Medical Centre (KCMC) and/or Mawenzi Hospital and receiving ART
* if > or =l to 18 years, able to understand the project and provide written, informed consent
* if < 18 years, a parent or guardian must provide written permission and participant must be able to assent
* all adolescents must also commit to attending 10 weekly CBT (SYV) sessions and 2 individual sessions.

Exclusion Criteria:

* Active psychosis, developmental delay, or cognitive disability that precludes active participation in consent process, intervention, and assessment interviews.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Participant attendance | weekly for 16 weeks during each intervention wave (over 2 years)
  Measure the percentage of participants who complete all intervention sessions and ability to interview participants for outcome measures over time.
Caregiver participation as measured by questionnaire | during 2 caregiver sessions
  Record willingness of caregivers to participate (if unwilling, why not) and attendance.
Caregiver participation as measured by attendance sheet | during 2 caregiver sessions
Fidelity as measured by weekly supervisor meeting | weekly for 16 weeks during the intervention wave (over 2 years)
Fidelity as measured by fidelity checklists | weekly for 16 weeks during the intervention wave (over 2 years)

SECONDARY OUTCOMES:
Change in Mental Health | pre-intervention, within 1 month post-intervention, 6- and 12- months post-intervention
  Compare the change in standard deviation of mental health symptoms on the PHQ-9, between the intervention group versus SOC.
Change in Mental Health | pre-intervention, within 1 month post-intervention, 6- and 12- months post-intervention
  Compare the change in standard deviation of mental health symptoms on the SDQ, between the intervention group versus SOC.
Change in Mental Health | pre-intervention, within 1 month post-intervention, 6- and 12- months post-intervention
  Compare the change in standard deviation of mental health symptoms on the UCLA PTSD-RI, between the intervention group versus SOC.
Change in ART adherence | pre-intervention, within 1 month post-intervention, 6- and 12- months post-intervention
  Compare the change in self-report adherence between the intervention group versus SOC.
Change in virologic outcomes | pre-intervention, within 1 month post-intervention, 6- and 12- months post-intervention
  Describe the proportion of youth with viral suppression (HIV-1 RNA < 400 copies/ml) in the intervention group and SOC.
Compare method of adherence measurement | pre-intervention, within 1 month post-intervention, 6- and 12- months post-intervention
  Compare self-report ART adherence with drug level concentration of hair samples.
Change in mental health (individual) | baseline to post-intervention, 6-, 12-,18- and 24-months
  Compare the change in standard deviation of mental health symptoms on the PHQ-9, SDQ, UCLA PTSD-RI at the individual level.
Change in adherence (individual) | baseline to post-intervention, 6-, 12-, and 24-months
  Compare the change in self-reported adherence and antiretroviral drug concentration in hair.
Change in HIV viral load (individual) | baseline to post-intervention, 6-, 12-, and 24-months
  Compare the change in HIV viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy E Dow, MD, MSc-GH, Principal Investigator — Duke University
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dow DE, Turner EL, Shayo AM, Mmbaga B, Cunningham CK, O'Donnell K. Evaluating mental health difficulties and associated outcomes among HIV-positive adolescents in Tanzania. AIDS Care. 2016 Jul;28(7):825-33. doi: 10.1080/09540121.2016.1139043. Epub 2016 Feb 3. PMID 26837437
- [Background] Ramaiya MK, Sullivan KA, O' Donnell K, Cunningham CK, Shayo AM, Mmbaga BT, Dow DE. A Qualitative Exploration of the Mental Health and Psychosocial Contexts of HIV-Positive Adolescents in Tanzania. PLoS One. 2016 Nov 16;11(11):e0165936. doi: 10.1371/journal.pone.0165936. eCollection 2016. PMID 27851797
- [Background] Gichane MW, Sullivan KA, Shayo AM, Mmbaga BT, O' Donnell K, Cunningham CK, Dow DE. Caregiver role in HIV medication adherence among HIV-infected orphans in Tanzania. AIDS Care. 2018 Jun;30(6):701-705. doi: 10.1080/09540121.2017.1391986. Epub 2017 Oct 23. PMID 29058461
- [Derived] Dow DE, Mmbaga BT, Gallis JA, Turner EL, Gandhi M, Cunningham CK, O'Donnell KE. A group-based mental health intervention for young people living with HIV in Tanzania: results of a pilot individually randomized group treatment trial. BMC Public Health. 2020 Sep 4;20(1):1358. doi: 10.1186/s12889-020-09380-3. PMID 32887558

DOCUMENTS (1):
  • Informed Consent Form (2015-02-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT02888288/ICF_000.pdf